CLINICAL TRIAL: NCT01598155
Title: The Effect of Supragingival Biofilm Control, and the Combination of Supra and Subgingival Biofilm Control in Periodontal Health of Patients Participating in a Periodontal Preventive Maintenance Program - A Randomized Clinical Trial.
Brief Title: Effect of Supragingival Control Versus Supra- and Subgingival Control in the Periodontal Health During the Maintenance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Sabrina Carvalho Gomes, DDS, PhD, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGomes 01
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Periodontitis
Keywords: dental biofilm; periodontitis; maintenance; randomized clinical trial; biomarkers; bacterias; gingival crevicular fluid
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supragingival biofilm control (Experimental)
  Interventions: Procedure: Group 1 - Supragingival biofilm control
- Supra- and subgingival biofilm control (Experimental)
  Interventions: Procedure: Group 2 - Supra- and subgingival biofilm control

INTERVENTIONS:
Procedure: Group 1 - Supragingival biofilm control — 30 days after the end of periodontal treatment, participants assigned to this group, will receive every 3 months (over 24 months):
  * Scaling, planning and polishing coronary surface;
  * Education and motivation for oral hygiene and daily supragingival biofilm control by the patient.
  Other Names: G1
  Arms: Supragingival biofilm control
Procedure: Group 2 - Supra- and subgingival biofilm control — 30 days after the end of periodontal treatment, participants assigned to this group, will receive every 3 months (over 24 months):
  * Scaling, planning and polishing of coronary surface;
  * Education and motivation for oral hygiene and daily supragingival biofilm control by the patient;
  * Subgingival scaling and root planning in sites with persistent bleeding on probing and probing depth unchanged.
  Other Names: G2
  Arms: Supra- and subgingival biofilm control

SUMMARY:
Seventy patients will be previously treated for moderate-to-severe periodontitis according to their individual needs. Thirty days after completion of periodontal treatment, these patients will be randomized to one of the following groups of periodic preventive maintenance (PPM): G1 - performed only control supragingival; G2 - performed supra and subgingival control (when necessary).

The maintenance consultations will be scheduled every 3 months for 24 months. The hypothesis is that the effect of the supragingival control (conducted over 24 months) will be similar to the effect of the supra- and subgingival control combined, above the restoration and progression of periodontitis.

DETAILED DESCRIPTION:
This randomized clinical trial, single-blind, aims to compare the effect of the supragingival biofilm control with the effect of supra- and subgingival biofilm control, performed by the patient-professional binomial, in periodontal patients treated, above the restoration and progression of periodontitis during the preventive periodic maintenance (PPM). Seventy patients with moderate-to-severe periodontitis, aged from 35 years, will be included. Participants will be periodontally treated according to their needs. After 30 days of the end of treatment, participants will be randomized (stratified for smoking) in two groups: Group 1 (G1)- Supragingival biofilm control; Group 2 (G2)- Supra and subgingival biofilm control. MPP consultation will take place every 3 months, for 24 months, in which the G1 will only receive procedures of supragingival biofilm control, and G2 will receive, beyond the supragingival control, subgingival interventions.

ELIGIBILITY:
Inclusion Criteria:

* age from 35 years;
* present at least 12 teeth in the mouth;
* patients diagnosed with moderate-to-severe periodontitis according to the criteria of the AAP (1999):

  * to present ≥ 2 interproximal sites with AL ≥ 6 mm AND ≥1 interproximal site with PD ≥ 5 mm; or
  * to present ≥ 2 interproximal sites with AL ≥ 3mm OR ≥ 2 interproximal sites with PD ≥ 5 mm (in different teeth).

Exclusion Criteria:

* presence of systemic conditions unfavorable to periodontal treatment (diabetes, cardiovascular changes with antimicrobial prophylaxis indicated);
* positive history of periodontal treatment and maintenance in the 12 months preceding the study;
* positive history of using anti-inflammatory drugs and antibiotics in the 3 months prior to initial consultation;
* patients in use of fixed orthodontic appliance;
* pregnant patients.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Mean Attachment Loss (AL) | 24 months
  AL: defined as the distance from the CEJ to the bottom of the pocket/sulcus.

SECONDARY OUTCOMES:
Periodontal Probing Depth (PPD) | 24 months
  PPD: defined as the distance from the free gingival margin to the bottom of the pocket/sulcus.
Microbiological markers | 24 months
  To assess the prevalence of P gingivalis, P micra and D pneumosintis on the subgingival plaque samples

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Carvalho Gomes, DDS, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- School of Dentistry, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Angst PDM, Van der Velden U, Susin C, Gomes SC. Supportive periodontal care with or without subgingival instrumentation: Microbiological results of a 2-year randomized clinical trial. J Clin Periodontol. 2024 Oct;51(10):1302-1310. doi: 10.1111/jcpe.14038. Epub 2024 Jul 2. PMID 38956881
- [Derived] Mendez M, Angst PDM, Oppermann RV, van der Velden U, Gomes SC. Oral health-related quality of life during supportive periodontal therapy: results from a randomized clinical trial. J Clin Periodontol. 2021 Aug;48(8):1103-1110. doi: 10.1111/jcpe.13473. Epub 2021 Jun 17. PMID 33899268
- [Derived] Angst PDM, Finger Stadler A, Mendez M, Oppermann RV, van der Velden U, Gomes SC. Supportive periodontal therapy in moderate-to-severe periodontitis patients: A two-year randomized clinical trial. J Clin Periodontol. 2019 Nov;46(11):1083-1093. doi: 10.1111/jcpe.13178. Epub 2019 Sep 2. PMID 31378975